CLINICAL TRIAL: NCT00816101
Title: Efficacy of the PROCELLERA™ Wound Dressing in the Healing of Wounds After a Curettage and Electrodesiccation of Skin Lesions
Brief Title: Efficacy Study of a New Antimicrobial Wound Dressing to Treat Wounds Caused by Curettage and Electrodesiccation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vomaris Innovations (Industry)
Responsible Party: Manager of Clinical Affairs, Vomaris Innovations, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XSMP-002
Record Dates: First submitted 2008-10-21; First posted 2008-12-31 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Acute Wounds
Keywords: Curettage and electrodesiccation; acute wounds; partial thickness wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PROCELLERA™Antimicrobial Dressing (Experimental): Dressing changes every 3 days, more frequently if needed
  Interventions: Other: Procellera™ Antimicrobial Dressing
- Mepilex® Border Lite (Active Comparator): Dressing changes every 2-3 days, more frequently if needed
  Interventions: Other: Mepilex® Border Lite
- Band-Aid® Adhesive Bandage (Active Comparator): Dressing changes every 2-3 days, more frequently if needed.
  Interventions: Device: Adhesive Bandage

INTERVENTIONS:
Other: Procellera™ Antimicrobial Dressing — Dressing indicated for partial and full-thickness wounds.
  Other Names: PROCELLERA™; Prosit™ Antimicrobial Dressing; Prosit™ Technology
  Arms: PROCELLERA™Antimicrobial Dressing
Other: Mepilex® Border Lite — Self-adherent foam dressing
  Other Names: Mepilex®
  Arms: Mepilex® Border Lite
Device: Adhesive Bandage — Adhesive bandage
  Other Names: Band-Aid® Adhesive Bandage
  Arms: Band-Aid® Adhesive Bandage

SUMMARY:
The purpose of this pilot clinical study is to compare healing rates, pain levels, and incidence of wound complications including infection with the use of a moist PROCELLERA™ Antimicrobial Wound Dressing when compared to a standard dressing, Mepilex® Border Lite, following curettage and electrodesiccation of skin lesions.

ELIGIBILITY:
Inclusion Criteria:

If female, must either be not of childbearing potential or if they are of childbearing potential must have a negative urine pregnancy test.

* Wound size greater than 1x1 cm
* Wounds must be ≥5 cm away from all other wounds
* Wound size must not be diminished in size greater than 10% between enrollment in study and the prescreening
* Participant agrees to participate in follow-up evaluation
* Participant must be able to read and understand informed consent, and sign the informed consent

Exclusion Criteria:

* Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study
* Participant is to receive another topical antimicrobial agent other than the study dressing
* Participant with sensitivity or adverse reactions to silver or zinc
* Pregnancy or nursing an infant or child
* Immunosuppression
* Active or systemic infection
* Peripheral vascular occlusive disease
* Collagen vascular disease
* Connective tissue disease
* Diabetes
* Venous stasis ulcers
* Participant undergoing active cancer chemotherapy
* Chronic steroid use
* Decision impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott N Sheftel, MD, Principal Investigator — Sheftel Associates Dermatology
Locations (1):
- Sheftel Associates Dermatology, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: June 2008-August 2008 Location: Dermatology Clinic
Groups:
- Procellera Dressing: Antimicrobial dressing for partial and full-thickness wounds. Produces small amount of current when in contact with conductive fluid. Used as primary contact layer for wound following curettage and electrodesiccation.
  Dressing changes every 3 days, more frequently if needed
- Mepilex® Border Lite: Self-adherent soft silicone foam dressing. Placed over wound following curettage and electrodesiccation. Dressing changes every 2-3 days, more frequently if needed
- Band-Aid® Adhesive Bandage: Adhesive bandage containing absorbtive pad secured to self-adherent strip. Placed over wound caused by curettage & electrodesiccation. Dressing changes every 2-3 days, more frequently if needed.
Period: Overall Study
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage
Started | 13 | 8 | 5
Completed | 13 | 8 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage | Total
Number analyzed (Participants) | 13 | 8 | 5 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 12 | 7 | 4 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 76.6 (8.4) | 74.8 (9.9) | 76.6 (8.4) | 74.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 8
  Male | 9 | 6 | 3 | 18
Region of Enrollment [Number; unit: participants]
  United States | 13 | 8 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced 50% or Greater Wound Healing
Description: Participants were assessed to see whether or not the wound area was reduced by at least 50%, and the number of such participants is reported
Time Frame: 3 Weeks
Measure: Number; unit: Participants
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage
Number analyzed (Participants) | 13 | 8 | 5
Participants | 13 | 7 | 4

2. Secondary Outcome: Number of Patients Reporting Pain
Description: Participants recorded their subjective pain level on a 0-10 Numeric Pain Chart 3x/day (0=no pain, 10=worst pain imaginable), until they had no pain for 3 consecutive days. Participants were also given a Patient Medication Log to complete at home to record RX and OTC medication they took to relieve pain. They were instructed to write the medication name, dosage, and amount of pills they took, as well as time taken, every day they took pain medication. Participants reporting pain had an associated score.
Time Frame: 3 Weeks
Measure: Number; unit: Participants
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage
Number analyzed (Participants) | 13 | 8 | 5
Participants | 0 | 0 | 0

3. Secondary Outcome: Erythema at Week 3
Description: At each weekly follow up visit, wound erythema was evaluated by the clinician on a scale of 0-4, with "0" being "No erythema", "1" being "Very slight erythema", "2" being "Well defined erythema", "3" being "Moderate to severe erythema" and 4 being "Severe erythema to slight eschar formation"
Time Frame: 3 Weeks
Measure: Mean (Standard Deviation); unit: Erythema Scores on a Scale
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage
Number analyzed (Participants) | 13 | 8 | 5
Erythema Scores on a Scale | 0.45 (0.82) | 1.29 (1.11) | 0.60 (0.55)

ADVERSE EVENTS:
Arm/Group | Procellera Dressing | Mepilex® Border Lite | Band-Aid® Adhesive Bandage
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No